CLINICAL TRIAL: NCT01648595
Title: Principal Investigator
Brief Title: Effect of Fentanyl on Pain Severity and Duration of Labor
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nahid Jahani Shoorab, Faculty of Midwifery, Mashhad University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Effect of Fentanyl
Record Dates: First submitted 2012-07-17; First posted 2012-07-24 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2006-01

CONDITIONS: Decrease Labor Pain
Keywords: Fentanyl; analgesia; duration of the active phase; pain severity
MeSH Terms: conditions — Agnosia; Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl (Experimental): In case group, 50 micrograms fentanyl was prescribed in two doses with an interval of 1 hour. In control group was not intervention.
  Interventions: Drug: Fentanyl
- Without Fentanyl (No Intervention): The control group did not receive Fentanyl.

INTERVENTIONS:
Drug: Fentanyl — In case group, 50 micrograms fentanyl was prescribed in two doses with an interval of 1 hour after being diluted in 4 cc normal saline
  Arms: Fentanyl

SUMMARY:
Background: There are two methods of pharmacologic and non- pharmacologic for reducing pain of delivery. It is necessary to be known effect of these drugs on the mother and fetus during labor adverse. Therefore, the purpose of this study was determination of effect of Fentanyl intravenously on pain severity during the active phase of labor.

ELIGIBILITY:
Inclusion Criteria:

* multiparas pregnant women (gravid 2-7),
* term singleton pregnancy,
* cephalic presentation,
* low risk pregnancy with no history of drug tolerance (addiction),
* medical and mental diseases.

Exclusion Criteria:

* Respiratory rate ≤ 8 or maternal bradycardia (pulse rate less than 60).

Ages: 21 Years to 37 Years | Sex: Female
Age Groups: Adult
Enrollment: 70
Dates: Start 2006-01; Primary Completion 2006-08; Study Completion 2006-09

PRIMARY OUTCOMES:
decrease pain and duration of the active phase considerably. | up to 8 months